CLINICAL TRIAL: NCT06986083
Title: A Randomized Controlled Trial of Modifications to Prostate Needle-Based Procedures
Brief Title: A Study of Changes to Prostate Procedures
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 25-085
Record Dates: First submitted 2025-05-20; First posted 2025-05-22 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: Needle-Based Procedures; IV sedation; Local anesthesia; 25-085
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: This is an ongoing, rolling phase III study. This is a surgical trial. Any agents administered to patients during the trial are part of routine care.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- No Local anesthesia (Experimental): No local anesthesia during transperineal biopsy under IV sedation
  Interventions: Procedure: Prostate Biopsy
- Local anesthesia (Active Comparator): Local anesthesia during transperineal biopsy under IV sedation
  Interventions: Procedure: Prostate Biopsy; Drug: Local anesthesia

INTERVENTIONS:
Procedure: Prostate Biopsy — Transperineal prostate biopsy
Drug: Local anesthesia — Local anesthesia in addition to IV sedation
  Arms: Local anesthesia

SUMMARY:
The purpose of this study is to look whether using local anesthesia during a transperineal prostate biopsy, while put to sleep by IV sedation, helps reduce the number of people who feel significant pain in the recovery room. The researchers will also look at how local anesthesia affects the amount of pain medication used, how quickly people can go home after the biopsy, and how well they recover after leaving the hospital.

ELIGIBILITY:
Inclusion Criteria:

Local anesthesia versus no local anesthesia during transperineal biopsy, while the patient is under IV sedation:

* Patients scheduled for transperineal prostate biopsy at the JRSC or Monmouth.

Standardization of a periprocedural pathway versus usual care for focal gland ablation:

* Patients scheduled for a partial prostate gland ablation procedure at the JRSC.

Exclusion Criteria:

Local anesthesia versus no local anesthesia during transperineal biopsy, while patient is under IV sedation:

* None

Standardization of a periprocedural pathway versus usual care for focal gland ablation:

* None

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate Cancer
Enrollment: 800 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Change in the proportion of patients experiencing significant pain | up to 1 day
  defined as at least one pain score ≥ 5 on a 0 - 10 scale in the post anesthesia care unit (PACU)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Fainberg, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org